CLINICAL TRIAL: NCT01862679
Title: Single Blind, Prospective, Randomised Comparative Study of High-flux Haemodialysis and Haemodiafiltration
Brief Title: Randomised Study of High-flux Haemodialysis and Haemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GN12RE153
Record Dates: First submitted 2013-04-22; First posted 2013-05-24 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hemodiafiltration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8 weeks HF haemodialysis / 8 weeks HD-filtration (Experimental): 8 weeks high-flux haemodialysis followed by 8 weeks haemodiafiltration
  Interventions: Other: High-flux haemodialysis; Procedure: Haemodiafiltration
- 8 weeks HD-filtration /8 weeks HF haemodialysis (Experimental): 8 weeks haemodiafiltration followed by 8 weeks high-flux haemodialysis
  Interventions: Other: High-flux haemodialysis; Procedure: Haemodiafiltration

INTERVENTIONS:
Other: High-flux haemodialysis — High-flux haemodialysis is the standard dialysis modality currently in use in the UK
Procedure: Haemodiafiltration — During Haemodiafiltration, the dialysis machine removes more water from the blood than during "normal" hemodialysis. The additional liquid is continually replaced with an ultra-pure solution. Thus, the machine exchanges a high volume of fluid during treatment and removes the liquid together with toxins from the blood.

SUMMARY:
The most common forms of renal replacement therapy currently in use are high flux haemodialysis (HF-HD) and haemodiafiltration (HDF). Although these techniques appear similar to the patient, there are important differences in what happens to the blood as it travels through the dialysis machine.

During HDF, the machine controls hydrostatic pressure across the dialyser to remove additional water together with toxins from the blood and this fluid volume is continually replaced with an ultra-pure solution. HDF has a theoretical advantage removing more waste substances, especially larger molecules, from the blood than HF-HD which may be of benefit to the patient in the medium to long term.Despite the theoretical advantages, trials have so far been unable to find any significant difference in death rates or the development of health problems among patients on HDF or HF-HD.

It is therefore important to examine other factors which may help doctors and patients to decide which treatment to use. The investigators have designed a study which aims to answer three main questions:

1. Does HDF make patients feel better?
2. Is blood pressure more stable on HDF in comparison with HF-HD?
3. Are Phosphate levels and other blood parameters better controlled with HDF than HF-HD?

The investigators will do this by randomly assigning patients on HF-HD to receive 2 months of either HF-HD or HDF with as equivalent treatment prescriptions as possible and without the patient knowing which treatment they are receiving. After two months the patients will switch to the alternative form of dialysis for a further two months. During the study the investigators will ask the patients how long it took them to recover from the preceding session of dialysis, assess the frequency of symptomatic low blood pressure and also perform blood tests at set intervals to measure specific blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* Receiving HF-HD for at least 3 months
* Reliable vascular access (i.e. use of the same fistula, graft or tunnelled central venous catheter for at least 1 month)
* Aged 18 or older

Exclusion Criteria:

* Currently receiving HDF
* Emergency hospital admissions within the preceding 4 weeks
* Life expectancy less than 6 months
* Neoplasia
* Unable to give informed consent
* Unable to perform QoL questionnaire or self report recovery post-dialysis time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in the average time taken to fully recover post dialysis | Baseline compared 8 week treatment point
  Self-assessment by patient of hours/mins to full recovery after dialysis

SECONDARY OUTCOMES:
Number of symptomatic hypotension events | Number of events noted by nurse at each dialysis session in each of the two arms of the study. Each arm= 3 sessions per week for 8 weeks
Number of dialysis circuit clotting events | Number of events noted by nurse at each dialysis session in each of the two arms of the study. Each arm= 3 sessions per week for 8 weeks
Pre-dialysis serum concentrations of potassium | Measured at baseline, and after 4 and 8 weeks of each treatment period
Pre-dialysis serum concentrations of phosphate | Measured at baseline, and after 4 and 8 weeks of each treatment period
Pre-dialysis serum concentrations of vitamin B12. | Measured at baseline, and after 4 and 8 weeks of each treatment period
Pre-dialysis serum concentrations of PTH. | Measured at baseline, and after 4 and 8 weeks of each treatment period
Pre-dialysis serum concentrations of beta-2-microglobulin | Measured at baseline, and after 4 and 8 weeks of each treatment period
Pre-dialysis serum concentrations of betaine | Measured at baseline, and after 4 and 8 weeks of each treatment period
Pre-dialysis serum concentrations of interleukin-6 | Measured at baseline, and after 4 and 8 weeks of each treatment period
Kt/V urea. | : Measured at baseline, and after 4 and 8 weeks of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Robert MacTier, Md, FRCP, Study Director — NHS Greater Glasgow and Clyde
Locations (1):
- NHS Greater Glasgow andClyde, Glasgow, United Kingdom